CLINICAL TRIAL: NCT07322211
Title: A Study to Evaluate the Clinical Performance and Safety of UNICON Silicone Hydrogel Daily Disposable Soft Contact Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unicon Optical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNC-002
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Refractive Ametropia
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label, single-arm, dispensing study. (Experimental): Qualis (linofilcon A) Soft (Hydrophilic) Daily Disposable Contact Lens
  Interventions: Device: Treatment

INTERVENTIONS:
Device: Treatment — Test lenses will be worn on a daily disposable basis for up to 13 weeks. Subjects will be instructed to wear the test lenses at least 6 hours a day, a minimum of 5 days per week.

SUMMARY:
13 weeks, open-label, daily disposable contact lens dispensing study.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the safety and clinical performance of the investigational soft contact lens when worn in a daily wear modality, by assessing total suspended eye(s) as the primary variable.

ELIGIBILITY:
Inclusion Criteria:

1. Adult with an age ≥ 18;
2. Be a currently adapted soft contact lens wearer who successful wear of soft contact lenses in both eyes for a minimum of 5 days per week and 6 hours per day within 3 months prior to study screening (by verbal confirmation);
3. Participant must be stop wearing any contact lenses more than 7 days prior to screening;
4. Able to wear contact lenses within a range of power from -2.00D to -6.00D (0.25 D steps) in both eyes;
5. Astigmatism of 1.25D or less in both eyes;
6. Be correctable to a visual acuity of 1.0 decimal (0.0 logMAR) or better in each eye;
7. Participant must be able to be successfully fit with study lenses;
8. The participant must appear able and willing to adhere to the instructions set forth in this clinical protocol;
9. The participant must read and sign the Informed Consent Form.

Exclusion Criteria:

1. Women who are currently pregnant;
2. Women who are lactating or planning a pregnancy at the time of enrollment (by verbal confirmation at the screening visit);
3. Any use of systemic or ocular medications (e.g., non-steroidal anti-inflammatory eye drops, ophthalmic steroids) within 30 days prior to study enrollment for which contact lens wear could be contraindicated, as determined by the investigator;
4. Any current or history ocular or systemic disease which may interfere with contact lens wear, as determined by the investigator;
5. Any current or previous orthokeratology treatment within 90 days prior to study enrollment, or planned for orthokeratology treatment during the study;
6. Any previous history of ocular and/or refractive surgery (e.g., radial keratotomy, PRK, LASIK, etc.) or planned for ocular and/or refractive surgery during the study;
7. Current or history of herpetic keratitis in either eye;
8. Current or history of intolerance, hypersensitivity or allergy to silicone hydrogel soft contact lenses or any component of the study products;
9. Current clinical finding of entropion, ectropion, chalazia, recurrent styes, glaucoma, pathologically dry eye (defined as Schirmer test < 5 mm/5 min), recurrent corneal erosions, aphakia, or moderate or above corneal distortion;
10. Employee of Department of Ophthalmology and clinic (e.g., Investigator, Coordinator, Technician);
11. Participation in any interventional clinical trial within 30 days prior to study enrollment;
12. Any biomicroscopy findings at screening that are Grade 3 or higher and/or corneal neovascularization that is Grade 2 or higher and/or presence of corneal infiltrates;
13. Any history of a contact lens-related corneal inflammatory or infectious event within 12 months prior to study enrollment that may contraindicate contact lens wear;
14. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator;
15. Participants are considered ineligible for the study as judged by the investigator.

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Total suspended eye(s) | From enrollment to the end of treatment at 13 weeks
  To evaluate the safety of study lenses by the total suspended eye(s) occurrence rate during the study period.

SECONDARY OUTCOMES:
Tabulation of Discontinued Eye(s) | From enrollment to the end of treatment at 13 weeks
  A tabulation of eyes discontinued from the study with reasons and the safety evaluation of the investigational lens evaluated based on these eye(s).
Tabulation of Subjective Symptoms | From enrollment to the end of treatment at 13 weeks
  Participant's symptoms, problems, and complaints will be collected via questionnaires and interviews at each visit. A tabulation of reported subjective symptoms will be compiled by visit and incidence rate, and the safety of the investigational lens will be evaluated accordingly.
Tabulation of Slit-Lamp Microscopy Findings | From enrollment to the end of treatment at 13 weeks
  Anterior segment findings observed during slit-lamp examination will be assessed according to the Slit-Lamp Examination Criteria (Appendix 1). A tabulation of slit lamp findings by visit, eyes and incidence rate will be created, and the safety of the investigational lens will be evaluated based on these findings.
Tabulation of Adverse Event(s) | From enrollment to the end of treatment at 13 weeks
  A tabulation of adverse event(s) (AEs) and serious adverse event(s) (SAEs) occurring during the study period will be created, and an assessment of the safety of the investigational lens will be conducted.
Tabulation of Adverse Device Effect(s) | From enrollment to the end of treatment at 13 weeks
  A tabulation of adverse device effect(s) (ADEs) and serious adverse device effects (SADEs) will be created. Calculate the incidence rates, and the safety of the investigational lens will be evaluated accordingly.
Tabulation of Device Deficiencies | From enrollment to the end of treatment at 13 weeks
  A tabulation of Device Deficiencies occurring during the trial will be compiled, and the safety of the investigational lens will be evaluated.
Contact Lens Corrected Visual Acuity | From enrollment to the end of treatment at 13 weeks
  The percentage of eyes achieving a lens-corrected visual acuity of ≥1.0 decimal (0.0 logMAR) at the final visit will be evaluated. If an eye does not achieve a visual acuity of 1.0 with the contact lens alone, but attains ≥1.0 after additional correction with spectacles, it shall be considered as meeting the 1.0 threshold.
Mean of Contact Lens Corrected Visual Acuity | From enrollment to the end of treatment at 13 weeks
  The mean of lens-corrected visual acuity (best corrected visual acuity while wearing the lenses) at the final examination will be calculated. The lower limit of the 95% confidence interval (95% CImin) will be statistically evaluated to confirm that it is ≥1.0.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
This study is intended for internal re-verification of the company's products and is not intended for external disclosure or use.

REFERENCES:
- [Background] WMA Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects. 75th WMA General Assembly, Helsinki, Finland, October 2024.
- [Background] ISO 14155:2020 Clinical investigation of medical devices for human subjects - Good clinical practice.
- [Background] ISO 11980:2012 Ophthalmic optics - Contact lenses and contact lens care products - Guidance for clinical investigations.
- [Background] Chalmers RL, Hickson-Curran SB, Keay L, Gleason WJ, Albright R. Rates of adverse events with hydrogel and silicone hydrogel daily disposable lenses in a large postmarket surveillance registry: the TEMPO Registry. Invest Ophthalmol Vis Sci. 2015 Jan 8;56(1):654-63. doi: 10.1167/iovs.14-15582. PMID 25574042
- [Background] Approaches to Clinical Evaluation of Standard Contact Lenses 標準的なコンタクトレンズの臨床評価に関する考え方 (Japan Independent Industry Guidelines 業界自主指針; August 1, 2009 平成21 年8 月1 日).